CLINICAL TRIAL: NCT05614843
Title: Pilot Study Evaluating the Impact of a Photobiomodulation Therapy on Xerostomia and Hyposalivation in Patients With Head and Neck Cancer Post-Radiotherapy
Brief Title: Photobiomodulation Therapy in Patients With Head and Neck Cancer Post-Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Noelia Galiano-Castillo, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBM_CANCER; PPJIA2020-15 (Other Grant/Funding Number: Universidad de Granada); PI-0187-2021 (Other Grant/Funding Number: Consejería de Salud y Familias (Junta de Andalucía))
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Xerostomia
Keywords: Quality of Life; Neoplasms; Xerostomia; Low-Level Light Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants who meet the inclusion and exclusion criteria will be randomized to one of the two study groups using a random number generation program (www.randomizer.org). The randomization sequence will be prepared by a member external to the investigation to respect the masking in terms of randomization of the participants, thus reducing the risk of bias during the evaluations. Therefore both patients and evaluator will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM group (Experimental): Energy density 7.5 J / cm2
  Interventions: Device: Energy density photobiomodulation (7.5)
- Control group (Placebo Comparator): The placebo control group will carry out the same protocol used in irradiated patients (including the use of protective goggles) using the same laser device to imitate a real irradiation; however, the device will be turned off and recording of the emission sounds will be used to give the patient the hearing sensation of the PBM therapy.
  Interventions: Device: Sham placebo

INTERVENTIONS:
Device: Energy density photobiomodulation (7.5) — A total of 22 points will be treated (extraoral and intraoral). 2 sessions per week, for 3 months (24 sessions in total).
  Arms: PBM group
Device: Sham placebo — A total of 22 points will be treated (extraoral and intraoral). 2 sessions per week, for 3 months (24 sessions in total).
  Arms: Control group

SUMMARY:
Patients with head and neck cancer post-radiotherapy may improve their perceived and amount of saliva after a 3-month Photobiomodulation (PBM) therapy focuses on three main salivary glands (parotid, submandibular and sublingual glands).

DETAILED DESCRIPTION:
The use of PBM therapy in survivors with head and neck cancer may be an effective treatment to improve xerostomia and hyposalivation as side effects of radiotherapy. Although there is some scientific evidence on its benefits during or after radiotherapy, it is not sufficient to establish it as an effective treatment. For these reasons, studies of higher methodological quality such as randomized controlled trials, are needed. This study aims to demonstrate the benefits of PBM therapy on xerostomia and hyposalivation in survivors with head and neck cancer undergone radiotherapy, and whether the effects are maintained after a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with head and neck cancer
* Persistent xerostomia after radiotherapy
* ≥18 years
* Irradiated with radiotherapy in the major salivary glands (parotid, submandibular and sublingual)
* Grade 3 for dry mouth in Common Terminology Criteria for Adverse Events, CTCAE (version 5.0)
* Have completed medical treatment with full response (complete remission) and receive medical clearance for participation.
* At least one month after radiotherapy completion, to reflect the possible presence of oral mucositis (sores) and/or radiodermatitis (inflammation) that limits adherence to treatment
* No use of drugs/devices/products (pilocarpine, cevimeline, amifostine, oral devices, humidifiers or herbs) to prevent or treat xerostomia before inclusion in the study, OR constant usage (do not change type and dosage) during 2 months before inclusion in the study

Exclusion Criteria:

* Relapse or metastasis
* Karnofsky activity scale <60
* Contraindications to PBM therapy (cardiac arrhythmias, pacemakers, photosensitivity, drugs with photosensitizing action, pregnancy)
* Patients with other comorbidities such as diabetes o polymedication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Xerostomia severity. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Xerostomia Inventory consists of 11 items, the total score ranges from 11 to 55 points, and represents the severity of chronic xerostomia. Higher scores mean a worse outcome.
Salivary flow rate. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Determines the amount of unstimulated saliva (ml) produced in 3 minutes. Higher amount means less hyposalivation.
General and specific quality of life in patients with head and neck cancer. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 assesses overall quality of life. It is a valid questionnaire and widely used in cancer population. High score for functional scales and global health status represents better outcomes. Higher symptom scales/items scores mean a worse outcome. In addition, its specific head and neck module (EORTC QLQ-H&N35) where higher symptom scales/items scores mean a worse outcome.
Nutritional and oral status. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Assesses through a Eating Assessment Tool questionnaire (EAT-10). Higher scores mean a worse outcome.
Maximum mouth opening. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Determine maximum mouth opening (mm) as the inter-incisor distance using a sliding caliper. More distance means better mobility.

SECONDARY OUTCOMES:
Pressure pain threshold. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Using a digital algometer in C5-C6 joint, upper trapezius, levator scapulae, masseter, temporalis, sternoclavicular joint and the tibialis anterior (distal point). Higher values mean higher pain pressure threshold.
Fitness Scale. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  The International Fitness Scale (IFIS) assesses overall fitness, cardio-respiratory, muscular, speed and flexibility dimensions using a 5-point Likert scale ('very poor', 'poor', 'average', 'good' and 'very good'). Higher scores mean a better outcome.
Mood status. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  The Spanish version of the Scale for Mood Assessment (EVEA) assesses mood state with a range of 0 to 10. It consists of 4 subscales: sadness-depression, anxiety, anger-hostility and happiness. Higher scores mean a worse outcome.
Quality of sleep. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  The Pittsburgh Sleep Quality Index will be used to evaluate the perceived quality of sleep in its Spanish version. Higher scores mean a worse outcome.
Physical activity level. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  The International Physical Activity Questionnaire (IPAQ-SF) is a tool that it will be used to evaluate physical activity. Different types of physical activities will be recorded (walking, moderate intensity activities, and vigorous intensity activities) during the last 7 days. More time means more amount of physical activity.
Functional capacity. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Using walked distance (m) during 6-minutes walking test. Longer distance means better outcome.
Risk of falls. | Change from Baseline to 12 weeks (after intervention) and to 6 months (follow-up).
  Using time (s) during Test Up and Go (TUG). Less time means less risk of falls.

OTHER OUTCOMES:
Safety and adverse events | 12 weeks (after intervention).
  Each adverse event is characterized by severity (grade 1 [mild] to 5 [death]), expectation (expected or unexpected) and potential relationship with participation in our study (unrelated, possibly related, or related to the study) using Common Terminology Criteria for adverse events (version 5.0). Higher scores mean a worse outcome.
Satisfaction questionnaire. | 12 weeks (after intervention).
  Each patient will mark his/her experience after PBM therapy. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia Galiano-Castillo, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences, Granada, Spain

REFERENCES:
- [Derived] Lopez-Garzon M, Plata-Peregrina MDC, Perez-Sanchez EI, Lozano-Lozano M, Artacho-Cordon F, Galiano-Castillo N. Photobiomodulation for restoring salivary flow after radiotherapy in head and neck cancer: a randomised placebo-controlled trial. BMC Oral Health. 2025 Sep 26;25(1):1468. doi: 10.1186/s12903-025-06735-3. PMID 41013422